CLINICAL TRIAL: NCT01604863
Title: Multi-Center, Open-Label Phase 1B Study to Evaluate the Safety and Tolerability of HGS1036 in Combination With Paclitaxel and Carboplatin, Cisplatin and Etoposide, or Docetaxel in Subjects With Advanced Solid Malignancies
Brief Title: A Study of HGS1036 in Combination With Chemotherapy in Subjects With Advanced Solid Malignancies
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Study suspended prior to enrollment
Sponsor: Human Genome Sciences Inc., a GSK Company (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGS1036-C1118
Record Dates: First submitted 2012-01-23; First posted 2012-05-24 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Cancer
Keywords: Solid Tumors; Cancer; Lung Cancer; Prostate Cancer; Mesothelioma; Small Cell lung Cancer
MeSH Terms: conditions — Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Mesothelioma; Small Cell Lung Carcinoma | interventions — Paclitaxel; Carboplatin; Cisplatin; Etoposide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (Experimental): HGS1036 + Paclitaxel + Carboplatin
  Interventions: Drug: HGS1036 + Paclitaxel + Carboplatin
- Arm B (Experimental): HGS1036 + Cisplatin + Etoposide
  Interventions: Drug: HGS1036 + Cisplatin + Etoposide
- Arm C (Experimental): HGS1036 + Docetaxel
  Interventions: Drug: HGS1036 + Docetaxel

INTERVENTIONS:
Drug: HGS1036 + Paclitaxel + Carboplatin — HGS1036 10 or 20 mg/kg, IV once weekly in each 21-day cycle. Paclitaxel 175 mg/m2 or 200 mg/m2, IV and carboplatin AUC 6.0 mg∙min/mL, IV every 3 weeks on Day 1 of each 21-day cycle.
  Arms: Arm A
Drug: HGS1036 + Cisplatin + Etoposide — HGS1036 10 or 20 mg/kg, IV once weekly in each 21-day cycle and cisplatin 60-80 mg/m2, IV on Day 1 and etoposide 100-120 mg/m2, IV on Days 1, 2, and 3 of each 21 day cycle.
  Arms: Arm B
Drug: HGS1036 + Docetaxel — HGS1036 10 or 20 mg/kg, IV once weekly in each 21-day cycle and docetaxel 75 mg/m2, IV on Day 1 of each 21-day cycle.
  Arms: Arm C

SUMMARY:
The primary purpose of this study is to determine the maximally tolerated dose (MTD) of HGS1036 when used in combination with the standard chemotherapeutic regimens paclitaxel plus carboplatin, cisplatin plus etoposide, or docetaxel.

DETAILED DESCRIPTION:
This study will consist of 3 regimens each containing 2 dose levels of HGS1036 and full dose chemotherapy. Patients will be treated in sequence with HGS1036 at planned dose levels of 10 mg/kg and 20 mg/kg. Patients who demonstrate stable disease or better may continue to receive HGS1036 until progressive disease, unacceptable toxicity, patient requests discontinuation of study treatment, or the Investigator feels further treatment is not in the patient's best interest. After discontinuation of HGS1036, subjects will be followed for 30 days after the last dose of HGS1036 for safety. The end of study will be defined as 1 year after the last subject begins treatment of HGS1036. Any subject still receiving HGS1036 at this pre-defined end of study, may continue to receive HGS1036, but the only study assessments required will be for safety.

ELIGIBILITY:
Inclusion Criteria:

* Have a histological or cytological diagnosis of malignant solid neoplasm requiring systemic chemotherapy.
* Age ≥18 years.
* ECOG performance status 0-1.
* Adequate organ function.
* Adequate hematological function.
* Have the ability to understand the requirements of the study, provide written informed consent, and comply with the study protocol procedures.
* Consent to collection of previously obtained, archival biopsy or surgical specimens of the currently treated malignancy when available.

Exclusion Criteria:

* Significant cardiac disease.
* Eye trauma or disease.
* Ocular surgery or blunt force trauma to the eye requiring treatment within 3 months prior to first dose of HGS1036.
* Presence or history of ≥ Grade 2 hemoptysis within 2 weeks of the first dose of HGS1036.
* Major surgery within 4 weeks of the first dose of HGS1036.
* Prior organ or allogeneic stem cell transplant.
* Non-healing or chronic wounds.
* Receipt of any anti-cancer therapy within 4 weeks prior to first dose of HGS1036.
* Receipt of any biological therapy (such as monoclonal antibodies) within 6 weeks of the first dose of HGS1036.
* Active CNS involvement by primary or metastatic tumor.
* Documented active infection requiring the use of systemic antibiotics.
* Pregnancy or lactation.
* Known HIV-positive serology, AIDS, or an AIDS-related illness.
* Conditions likely to increase the potential for abdominal perforation or fistula formation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Up to 1 year or longer if indicated.
Number of participants with adverse events | Up to 1 year or longer if indicated.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - Scottsdale, Arizona
  - Boston, Massachusetts